CLINICAL TRIAL: NCT04250805
Title: Trial Evaluating the Efficacy of the Combination of ROpivacaine With Reference XYlocaine in the Evaluation of Pain During the Installation of Percutaneous Radiological GASTrostomy
Acronym: GASTROXY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties in recruiting patients
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-1201; 2019-004835-22 (EudraCT Number)
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Cancer; Feeding Disorders
Keywords: Cancer; Gastrostomy; Percutaneous technique; Radiological guidance; Lidocaine; Ropivacaine; Pain
MeSH Terms: conditions — Neoplasms; Feeding and Eating Disorders; Pain | interventions — Lidocaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Active Comparator): Patients will receive Lidocaine alone during percutaneous gastrostomy under radiological guidance
  Interventions: Drug: Lidocaine
- Lidocaine and Ropivacaine (Experimental): Patients will receive Lidocaine and Ropivacaine during percutaneous gastrostomy under radiological guidance
  Interventions: Drug: Lidocaine; Drug: Ropivacaine

INTERVENTIONS:
Drug: Lidocaine — Patients will receive Lidocaine during percutaneous gastrostomy under radiological guidance.
Drug: Ropivacaine — Patients will receive Ropivacaine during percutaneous gastrostomy under radiological guidance.
  Arms: Lidocaine and Ropivacaine

SUMMARY:
Gastrostomy is an intra-gastric nutritional enteral device that could be put in place by percutaneous technique under radiological guidance: allowing local anesthesia. However, there is no clear recommendation about local analgesia during this exam. Operator can chose Lidocaine with a short period of action, or Ropivacaine with a longer period of action. The association of these two drugs could enhance the analgesia post procedure. The main objective of this study is to decrease maximal pain felt during a twenty four hour stay, after a gastrostomy under percutaneous technique with radiological guidance.

DETAILED DESCRIPTION:
Gastrostomy is an intra-gastric nutritional enteral device, allowing the nutritional support for patients presenting oral feeding disorders. Gastrostomy could be put in place by different manners:

* Chirurgical technique or endoscopy: with general anesthesia;
* Percutaneous technique under radiological guidance: allowing local anesthesia. This last one is better tolerated by weak patients, and involves less complication.

However, there is no clear recommendation about local analgesia during this exam. Operator can chose Lidocaine with a short period of action, or Ropivacaine with a longer period of action.

The association of these two drugs could enhance the analgesia post procedure. Indeed, pain felt during the twenty four hours post procedure seems to be the most frequent adverse effect reported by patients.

Pain could decrease significantly when Ropivacaine is added to the reference Xylocaine. Ropivacaine had already proved its efficacy in association with other antalgics.

The main objective of this study is to decrease maximal pain felt during a twenty four hour stay, after a gastrostomy under percutaneous technique with radiological guidance.

ELIGIBILITY:
Inclusion criteria :

* Major patient;
* Having an indication for placement of PRG (percutaneous radiological gastrostomy);
* Patient hospitalized for a minimum of 24 hours post gastrostomy;

Non-inclusion criteria :

* Pregnant or lactating woman;
* Legal incapacity or limited legal capacity. Medical or psychological conditions which do not allow the subject to understand the study and sign the consent (art. L.1121-6, L.1121-7, L.1211-8, L.1211-9);
* Not knowing how to read and / or write French;
* Allergy and / or known hypersensitivity to lidocaine and / or ropivacaine or to other local anesthetics with amide bond or to one of the excipients;
* Recurrent porphyrias (genetic, hereditary diseases affecting the production of hemoglobin);
* Patient on beta blockers during the installation of PRG (Percutaneous Radiological Gastrostomy);
* Indication of gastrostomy button placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Level of Pain | 24 hours
  Two points diminution for maximal pain felt during a twenty four hours after percutaneous gastrostomy under radiological guidance. It will be measured with a visual analogue scale starting at zero for no pain and ending at ten for maximal pain felt.

SECONDARY OUTCOMES:
Level of Anxiety and Depression | 10 days
  Hospital Anxiety and Depression scores will be reported and analysed for each patient. This scale is an instrument for detecting anxiety and depressive disorders. It has 14 listed items from 0 to 3. Seven questions relate to anxiety (total A) and seven others relate to the depressive dimension (total D), allowing thus obtaining two scores (maximum score of each score = 21). To detect anxious and depressive symptoms, the following interpretation can be offered for each of the scores (A and D):
  * 7 or less: absence of symptoms;
  * 8 to 10: doubtful symptomatology;
  * 11 and more: certain symptomatology.
Level of quality of life | 10 days
  Brief Pain Inventory scores will be reported to evaluate the level of the patients' quality of life. For each question, score is comprised between 0 and 10, with 0 meaning no pain or no resounding on life activity, and 10 meaning the worst pain ever, and the worst resounding on life activity.
Level of satisfaction | 10 days
  Patients' satisfaction about their analgesic care will be reported with a visual analogue scale starting at zero meaning no satisfaction, and ending at ten meaning the highest satisfaction possible.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Etievent, MD, Principal Investigator — Institut de Cancérologie Lucien Neuwirth
Locations (2):
- France (2):
  - CHU de Saint-Etienne, Saint-Priest-en-Jarez
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No